CLINICAL TRIAL: NCT02841150
Title: A Single-Dose, Open-Label, Randomized, Replicate Crossover Study in Healthy Adult Subjects to Assess the Bioequivalence of an Ibrutinib 560-mg Tablet Compared to the Four IMBRUVICA 140 mg Capsules
Brief Title: Study to Assess the Bioequivalence of Ibrutinib 560- Milligram (mg) Tablet to Four 140 -mg IMBRUVICA Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108171; 54179060CLL1021 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-06-15; First posted 2016-07-22 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Healthy
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Treatment Sequence 1 (Experimental): Participants will receive treatment A, on Day 1 of Intervention Period 1 followed by treatment B , on Day 1 of Intervention Period 2 followed by treatment A, Day 1 of Intervention Period 3 and then followed by treatment B, on Day 1 of Intervention Period 4. Each intervention Period will be separated by a washout period of 7-9 days.
  Interventions: Drug: IMBRUVICA (Treatment A); Drug: Ibrutinib (Treatment B)
- Treatment Sequence 2 (Experimental): Participants will receive treatment B, on Day 1 of Intervention Period 1 followed by treatment A, on Day 1 of Intervention Period 2 followed by treatment B, Day 1 of Intervention Period 3 and then followed by treatment A, on Day 1 of Intervention Period 4. Each intervention Period will be separated by a washout period of 7-9 days.
  Interventions: Drug: IMBRUVICA (Treatment A); Drug: Ibrutinib (Treatment B)

INTERVENTIONS:
Drug: IMBRUVICA (Treatment A) — IMBRUVICA (reference treatment), 4*140 milligram (mg), capsules.
  Other Names: Ibrutinib
Drug: Ibrutinib (Treatment B) — Ibrutinib (test treatment), 1*560 mg, tablet.

SUMMARY:
The purpose of this study is to demonstrate the bioequivalence (BE) of a new formulation of ibrutinib to the marketed Imbruvica formulation in healthy adults under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study, before any study related procedures take place
* Willing and able to adhere to the prohibitions and restrictions specified in the protocol
* If a woman, must be of non-childbearing potential, defined as either: a) Postmenopausal: A postmenopausal state is defined as no menses for at least 12 months without an alternative medical cause and a serum follicle stimulating hormone (FSH) level in the postmenopausal range (greater than [>]40 international units per liter [IU/L] or milliinternational units per milliliter [mIU/mL]). b) Permanently sterile: Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures (without reversal operation), bilateral oophorectomy, and/or transcervical sterilization
* If a woman, must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening and on Day -1 of each treatment period
* Non-smoker for at least 2 months prior to screening

Exclusion Criteria:

* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen/paracetamol, topical therapies, and hormone replacement therapy within 14 days before the first dose of the study drug is scheduled
* History of clinically significant allergies, especially known hypersensitivity or intolerance to sulfonamide or beta-lactam antibiotics
* Known allergy to the study drug or any of the excipients of the formulation
* Unable to swallow solid, oral dosage forms whole with the aid of water (participants may not chew, divide, dissolve, or crush the study drug)
* Positive test for human immunodeficiency virus type 1 (HIV-1) or HIV-2 antibodies at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Ibrutinib | Day 1 (Pre-dose) up to Day 3
  The Cmax is the maximum observed plasma concentration.
Time to reach maximum concentration (tmax) of Ibrutinib | Day 1 (Pre-dose) up to Day 3
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-last]) of Ibrutinib | Day 1 (Pre-dose) up to Day 3
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of Ibrutinib | Day 1 (Pre-dose) up to Day 3
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda[z]) of Ibrutinib | Day 1 (Pre-dose) up to Day 3
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Terminal Half-Life (t[1/2]) of Ibrutinib | Day 1 (Pre-dose) up to Day 3
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Maximum Plasma Concentration (Cmax) of IMBRUVICA | Day 1 (Pre-dose) up to Day 3
  The Cmax is the maximum observed plasma concentration.
Time to reach maximum concentration (tmax) of IMBRUVICA | Day 1 (Pre-dose) up to Day 3
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-last]) of IMBRUVICA | Day 1 (Pre-dose) up to Day 3
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of IMBRUVICA | Day 1 (Pre-dose) up to Day 3
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda[z]) of IMBRUVICA | Day 1 (Pre-dose) up to Day 3
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Terminal Half-Life (t[1/2]) of IMBRUVICA | Day 1 (Pre-dose) up to Day 3
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events as a measure of safety and tolerability | Baseline up to 14 days after last dose of study drug (Day 17)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States